CLINICAL TRIAL: NCT04784780
Title: Long-term Efficacy and Safety of Elobixibat for Chronic Constipation: a Multicenter, Randomised, Double-blind, Placebo-controlled Trial.
Brief Title: Long-term Elobixibat for Chronic Constipation
Acronym: TANK-27
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yokohama City University (Other)
Responsible Party: Principal Investigator, Takaomi Kessoku, Principal Investigator, Yokohama City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jRCTs031200363
Record Dates: First submitted 2021-02-28; First posted 2021-03-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Chronic Constipation
Keywords: Elobixibat; Chronic constipation; 12 week; Complete spontaneous bowel movement
MeSH Terms: interventions — elobixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elobixibat (Experimental): AJG533 (elobixibat) 10 mg orally once a day before meals for 12 weeks
  Interventions: Drug: Elobixibat 10mg
- Placebo (Placebo Comparator): AJG533 placebo orally once a day before meals for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elobixibat 10mg — Patients with chronic constipation are administered Elobixibat 10mg for 12 weeks
  Other Names: AJG533 10 mg
  Arms: Elobixibat
Drug: Placebo — Patients with chronic constipation are administered placebo for 12 weeks
  Other Names: AJG533 placebo
  Arms: Placebo

SUMMARY:
In this double-blind comparative study, AJG533 (elobixibat) 10 mg or AJG533 placebo was orally administered once daily before meals for 12 weeks in patients with chronic constipation, and the primary endpoint was the change from Week 2 of the observation period in the number of complete spontaneous bowel movements (CSBM) at Week 12 of the treatment period. The primary endpoint was the change in the number of complete spontaneous bowel movements (CSBM) from Week 2 of the observation period.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic constipation by the "Rome IV" criteria for chronic constipation
* Age: 20 years old or older and up to 85 years old (at the time of obtaining consent)
* Gender: any gender
* outpatients
* Patients who can obtain written consent
* Patients who can record their defecation, etc. in the patient's diary

At the time of allocation (dosing initiation criteria)

* Spontaneous bowel movements (SBM)* not more than 6 times during the 2-week observation period before the start of treatment
* Patients with no soft or watery stools (Bristol Stool Shape Scale 6 or 7) in spontaneous bowel movements during the 2-week observation period before the start of treatment.
* Patients who have not used concomitantly prohibited drugs or therapies during the observation period.

Exclusion Criteria:

* Patients with organic constipation or patients with suspected organic constipation.
* Patients with or suspected of having functional ileus.
* Patients with or suspected of having an inguinal hernia.
* Patients with a history of open surgery within 12 weeks before obtaining consent (excluding appendicitis resection).
* Patients with a history of surgical or endoscopic procedures related to cholecystectomy and papillotomy.
* Patients with complications of malignancy.
* Pregnant women, lactating women, women who may be currently pregnant, or patients who cannot consent to use contraception while participating in the study.
* Patients with serious renal, liver, or cardiac disease.
* Patients who are allergic to this study drug.
* Patients who have previously taken Goufis tablets (elobixibat).
* Patients with contraindications to rescue drugs (bisacodyl suppositories and prusenide tablets).
* Patients who are participating in another clinical study or who were participating in another clinical study within 4 weeks before consent was obtained, excluding observational studies.
* Patients who are judged by the principal investigator or sub-physician to be inappropriate for conducting this research.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the number of complete spontaneous bowel movements at week 12 | Week 12
  Change in the number of complete spontaneous bowel movements at week 12 of the treatment period from week 2 of the observation period. *Spontaneous defecation without residual sensation.

SECONDARY OUTCOMES:
Change in the number of complete spontaneous bowel movements in each week of the treatment period. | Each Week 1-11
  Change in the number of complete spontaneous bowel movements in each week of the treatment period.
Change in the number of spontaneous bowel movements in each week of the treatment. | Each Week 1-11
  Change in the number of spontaneous bowel movements in each week of the treatment.
Proportion of responders** in the number of SBMs during each week. | Each Week 1-11
  Proportion of responders** in the number of spontaneous bowel movements (SBMs) during each week of the treatment period.
  **In this study, we will investigate the effect of the treatment on the number of SBMs of a subject who has at least one more SBM per week than in the second week of the observation period, and at least three times per week.
Proportion of responders** in the number of CSBMs during each week. | Each Week 1-11
  Proportion of responders** in the number of complete spontaneous a bowel movements (CSBMs) during each week of the treatment period.
  **In this study, we will investigate the effect of the treatment on the number of CSBMs of a subject who has at least one more CSBMs per week than in the second week of the observation period, and at least three times per week.
The rate of a responder in the number of CSBM during the treatment period. | Week 12
  Definition of Responder: Patients with 3 or more CSBM per week and 1 or more CSBM per week from baseline for 9 weeks out of the entire treatment period (12 weeks), including at least 3 weeks in the treatment period weeks 9 to 12.
Percent change in fecal hardness based on the Bristol Stool Quality Scale at each week. | Each Week 1-11
  Percent change in fecal hardness from week 2 of the observation period based on the Bristol Stool Quality Scale at each week of the treatment period. the minimum is 1 and maximum values, is 7.Higher scores mean a better outcome.
The percentage of change in the presence or absence of residual sensation at each week. | Each Week 1-11
  The percentage of change from week 2 of the observation period in the presence or absence of residual sensation at each week of the treatment period.
Percent change in the degree of twitching at each week. | Each Week 1-11
  Percent change from week 2 of the observation period in the degree of twitching at each week of the treatment period.
The percentage of change in the presence or absence of bowel movements at each week. | Each Week 1-11
  The percentage of change in the presence or absence of bowel movements at each week of the treatment period from week 2 of the observation period.
Change in Japanese Patient assessment of constipation quality of life score | Week 4, 12
  Change in Japanese Patient assessment of constipation quality of life score at 4 and 12 weeks of the treatment period from the baseline (V2) of the study drug.the minimum is 0 and maximum values is 4.Lower scores mean a better outcome.
The changes in occupancy rate of intestinal microbiota. | Week 4, 12
  At 4 weeks and 12 weeks of the treatment period, the changes in occupancy rate of intestinal microbiota in feces from before the start of the study drug (V2) are examined.
The change in absolute values rates in blood and fecal bile acids. | Week 4, 12
  At 4 weeks and 12 weeks of the treatment period, the change in absolute values in blood and fecal bile acids from before the start of the study drug (V2) are examined.
The change in absolute values for organic acids. | Week 4, 12
  At 4 weeks and 12 weeks of the treatment period, the change in absolute values for organic acids in feces from before the start of the study drug (V2) are examined.
The change in absolute values of amino acids in blood and feces. | Week 4, 12
  At 4 weeks and 12 weeks of the treatment period, the change in absolute values of amino acids in blood and feces. from before the start of the study drug (V2) are examined.
The change in amount blood C4. | Week 4, 12
  At 4 weeks and 12 weeks of the treatment period, the change in amount blood C4 from before the start of the study drug (V2) are examined.

OTHER OUTCOMES:
Incidence of adverse events. | Each Week 1-11
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Takaomi Kessoku, M.D., PhD., Principal Investigator — Yokohama City University
Locations (1):
- Yokohama City University, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakajima A, Seki M, Taniguchi S, Ohta A, Gillberg PG, Mattsson JP, Camilleri M. Safety and efficacy of elobixibat for chronic constipation: results from a randomised, double-blind, placebo-controlled, phase 3 trial and an open-label, single-arm, phase 3 trial. Lancet Gastroenterol Hepatol. 2018 Aug;3(8):537-547. doi: 10.1016/S2468-1253(18)30123-7. Epub 2018 May 25. PMID 29805116
- [Derived] Tanaka K, Kessoku T, Yamamoto A, Takahashi K, Kasai Y, Ozaki A, Iwaki M, Kobayashi T, Yoshihara T, Misawa N, Kato T, Arimoto J, Fuyuki A, Sakai E, Higurashi T, Chiba H, Hosono K, Yoneda M, Iwasaki T, Kurihashi T, Nakatogawa M, Suzuki A, Taguri M, Oyamada S, Ariyoshi K, Kobayashi N, Ichikawa Y, Nakajima A. Rationale and design of a multicentre, 12-week, randomised, double-blind, placebo-controlled, parallel-group, investigator-initiated trial to investigate the efficacy and safety of elobixibat for chronic constipation. BMJ Open. 2022 May 30;12(5):e060704. doi: 10.1136/bmjopen-2021-060704. PMID 35636802